CLINICAL TRIAL: NCT00421083
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Assess Efficacy and Safety of Tadalafil (LY450190) in Subjects With Erectile Dysfunction Caused by Spinal Cord Injury
Brief Title: Efficacy and Safety of Tadalafil in Subjects With Erectile Dysfunction Caused by Spinal Cord Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9108; H6D-MC-LVFY
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Erectile Dysfunction; Spinal Cord Injuries
Keywords: Erectile dysfunction as a result of traumatic spinal cord injury
MeSH Terms: conditions — Erectile Dysfunction; Spinal Cord Injuries | interventions — Tadalafil

INTERVENTIONS:
Drug: tadalafil
  Other Names: LY450190; Cialis; IC351

SUMMARY:
This is a study of the efficacy and safety of on-demand dosing of tadalafil or placebo administered for 12 weeks to men with erectile dysfunction caused by spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* males who developed erectile dysfunction as a result of spinal cord injury. Injury must have occurred 6 months before the start of the study.
* at least 4 sexual intercourse attempts during the first 4 weeks of the study without medication assistance
* no use of other erectile dysfunction treatment for at least 4 weeks before receiving the first dose of study drug. Also cannot use any other erectile dysfunction treatment during the study.

Exclusion Criteria:

* Impotence caused by other primary sexual disorders including premature ejaculation or untreated endocrine diseases such as diabetes, hypopituitarism, hypothyroidism, or hypogonadism
* History of radical prostatectomy or other pelvic surgery with subsequent failure to achieve any erection and history of penile implant.
* History of cardiac conditions including angina requiring certain treatment with nitrates; heart disease or coronary conditions including myocardial infarction, bypass surgery, angioplasty or stent placement for a specified time before starting the study.
* Significant renal problems within 6 months before starting the study. Also, active liver disease including jaundice at beginning of study.
* History of other central nervous system injuries, other than spinal cord injury, 6 months before starting the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2004-09; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Safe and effective as shown by improvement on erectile function IIEF scores and SEP scores.

SECONDARY OUTCOMES:
Additional efficacy variables including GAQ, SEP, and IIEF subdomains. Quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com